CLINICAL TRIAL: NCT00689312
Title: Palatability of Oral Rehydration Solutions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stephen Freedman, Adjunct Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1000012122
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis
Keywords: Gastroenteritis; Pediatrics; Rehydration therapy
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Enfalyte
- 2 (Experimental)
  Interventions: Drug: Pediatric Electrolyte
- 3 (Experimental)
  Interventions: Drug: Pedialyte

INTERVENTIONS:
Drug: Enfalyte — Each patient will receive one 250 ml dose.
  Arms: 1
Drug: Pediatric Electrolyte — Each patient will receive one 250 ml dose.
  Arms: 2
Drug: Pedialyte — Each patient will receive one 250 ml dose.
  Arms: 3

SUMMARY:
The primary objective of this study is to compare the mean taste scores for three fruit flavored oral rehydration solutions in children aged 5-10 years old. The secondary objective is to compare the proportions of children who indicate a taste preference for one of the solutions.

DETAILED DESCRIPTION:
In Canada, acute gastroenteritis remains a major cause of morbidity and hospitalizations. This, in large part, is due to an inability to realize the full benefits of oral rehydration therapy. Because oral rehydration solutions have a salty taste, many mild to moderate dehydrated children refuse to drink them. This has resulted in pediatricians recommending inappropriate solutions and the unnecessary administration of intravenous fluids. Although two meta-analyses have concluded that rice-based ORS (Enfalyte) is as or more effective than traditional ORS in reducing stool output, the palatability of different oral rehydration solutions have never been evaluated.

This will be the first prospective trial comparing the palatability of the most commonly recommended oral rehydration solutions, Pedialyte and Enfalyte with a newer solution, Pediatric Electrolyte. Both Pedialyte and Pediatric Electrolyte contain sucralose, dextrose, and fructose while Enfalyte contains rice syrup solids. Although the latter is as, or more effective than Pedialyte in reducing stool output, palatability may limit its use. Taste is important as children with gastroenteritis are frequently nauseated and may refuse to drink or vomit when consuming less palatable solutions.

We hypothesize that, compared to children who receive a rice-based ORS (Enfalyte), those who receive a sucralose ORS (Pediatric Electrolyte or Pedialyte) will report a higher mean taste score, will prefer to drink the sucralose sweetened ORS if they had to consume a larger volume, and are more likely to drink the entire volume they are provided.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-10 years of age evaluated in The Hospital for Sick Children's emergency department

Exclusion Criteria:

* Children with diarrhea, a vomiting or diarrhea episode within 24 hours, head trauma, abdominal pain, upper respiratory symptoms, or nil per os status
* Patients with gastrointestinal symptoms

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Mean taste scores for Pedialyte, Pediatric Electrolyte, and Enfalyte. | Immediately following consumption of each solution.

SECONDARY OUTCOMES:
Proportions of children who indicate a taste preference for one of the solutions. | Immediately following consumption of each solution.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Freedman SB, Cho D, Boutis K, Stephens D, Schuh S. Assessing the palatability of oral rehydration solutions in school-aged children: a randomized crossover trial. Arch Pediatr Adolesc Med. 2010 Aug;164(8):696-702. doi: 10.1001/archpediatrics.2010.129. PMID 20679159